CLINICAL TRIAL: NCT05647330
Title: Phase II Clinical Study of Hydroxychloroquine Combined With Gemcitabine in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Hydroxychloroquine Combined With Gemcitabine in the Treatment of Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022213
Record Dates: First submitted 2022-09-15; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-09

CONDITIONS: Hydroxychloroquine; Gemcitabine; Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Gemcitabine; Chloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxychloroquine combined with gemcitabine (Experimental): 1. Hydroxychloroquine sulfate tablets: twice a day, each time (600mg). Continuous oral administration. Until the disease progresses or becomes intolerable.
  2. gemcitabine was administered intravenously at a dose of 1000mg/m2 for 30min,d1, 8, and every 3 weeks (21 days) until disease progression or intolerable toxicity, with a maximum duration of 2 years.
  Interventions: Drug: Hydroxychloroquine Combined With Gemcitabine

INTERVENTIONS:
Drug: Hydroxychloroquine Combined With Gemcitabine — Hydroxychloroquine combined with chemotherapy
  Other Names: chloroquine

SUMMARY:
To evaluate the efficacy and safety of hydroxychloroquine (600mgBID) combined with gemcitabine (1000mg/m2,d1,8) in the third-line and above treatment of advanced NSCLC.

DETAILED DESCRIPTION:
This study is a single-arm, open phase II prospective cohort study to evaluate the efficacy and safety of hydroxychloroquine (600mgBID) combined with gemcitabine in the treatment of advanced NSCLC patients with third-line and above treatment. After signing informed consent, the subjects were screened and eligible for inclusion in this study.

All enrolled subjects will be treated with (hydroxychloroquine 600mgBID) plus gemcitabine, and each patient will continue to receive the study drug until the end of the treatment cycle. The efficacy index and safety index were observed during the treatment.

1. Hydroxychloroquine sulfate tablets: twice a day, each time (600mg). Continuous oral administration. Until the disease progresses or becomes intolerable.
2. gemcitabine was administered intravenously at a dose of 1000mg/m2 for 30min,d1, 8, and every 3 weeks (21 days) until disease progression or intolerable toxicity, with a maximum duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven advanced lung squamous cell carcinoma or lung adenocarcinoma with negative EGFR and ALK gene mutations.
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, meaning that at least one lesion can be accurately measured by conventional techniques of CT or MRI.
* It is acceptable for patients who have received radiotherapy. It must be at least 4 months after radiotherapy, and all signs of toxicity must abate.
* The patient must be 18 years of age or above.
* The ECOG performance status of patients must be 0-1.
* Patients should not become pregnant or breastfeed because chemotherapy is considered to pose significant risks to the fetus/baby.
* The patient must have a life expectancy of more than three months.
* Patients must be able to understand and willing to sign written informed consent.
* Previously received systematic treatment with 2 regimens;
* Treatment with hydroxychloroquine sulfate tablets plus gemcitabine is required to be initiated within 28 days after informed consent;
* The function of vital organs should meet the following requirements as far as possible (if laboratory test values do not meet the following criteria, they can also be included in the registration after comprehensive evaluation by researchers) :

  1. Absolute neutrophil count ≥1.5×109/L;
  2. Platelets ≥80×109/L;
  3. Hemoglobin ≥9g/dL;
  4. Serum albumin ≥ 3G /dL;
  5. Total bilirubin ≤1.25×ULN;
  6. ALT and AST ≤2.5×ULN; If liver metastases were present, ALT and AST≤5×ULN;
  7. serum creatinine ≤1.25×ULN or creatinine clearance ≥50mL/min.

Exclusion Criteria:

* Patients with rapid progression after 1 or 2 cycles in first-line and second-line regimens.
* Persons with known allergies or metabolic disorders to any drug in the treatment regimen.
* Patients who had previously received hydroxychloroquine.
* Patients with known G6PD deficiency, severe psoriasis, porphyria, macular degeneration, or severe diabetic retinopathy were ineligible because of the potential for greater hydroxychloroquine toxicity.
* Symptomatic central nervous metastasis. Patients with asymptomatic brain metastases or stable brain metastases after treatment were eligible to participate in the study if they met all the following criteria: measurable lesions outside the central nervous system; No mesencephalon, pons, cerebellum, meninges, medulla oblongata or spinal cord metastases; Maintain clinical stability for at least 2 weeks.
* A history of psychotropic drug abuse, alcoholism or drug abuse;
* In the 6 months prior to study entry, the following conditions occurred: myocardial infarction, severe/unstable angina pectoris, New York Heart Association (NYHA) grade 2 or higher cardiac dysfunction, and poorly controlled arrhythmias (including QT c F interval men & GT; 450 m s, female & GT; 470 ms, QT cF interval calculated by Fridericia formula), symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism);
* Human immunodeficiency virus (HIV, HIV 1/2 antibody) positive; Acute or chronic active hepatitis B (HBsAg positive and HBV DNA & g t; 1*103/ml) or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA & g t; 15 iu/ml); Active pulmonary tuberculosis;
* Other factors that may affect patient safety or compliance as determined by the investigator. If there is a serious illness (including mental illness) that requires concomitant treatment, serious laboratory abnormalities, or other family or social factors.
* Patients deemed inappropriate for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 1years
  The proportion of patients whose tumor volume reduction reaches the predetermined value and can maintain the minimum time limit is the sum of the proportion of complete and partial remission.

SECONDARY OUTCOMES:
Disease control rate(DCR) | 2 years
  The percentage of patients with PR + Cr and SD after treatment in the number of evaluable cases, and the RECIST standard is at least 4 weeks
Progression-free survival(PFS) | 2 years
  The time between initiation of the study drug and the first recorded date of disease progression (PD) or death, depending on which occurred first. If no disease progression is observed, the cutoff date should be the date of the last tumor measurement.
Overall survival(OS) | 2 years
  The time from the beginning of treatment to (for any reason) death. The last follow-up time is usually calculated as the time of death for the subjects who have lost the visit before death

IPD SHARING:
Plan to Share IPD: No